CLINICAL TRIAL: NCT03318848
Title: Use of Bed Bath Video During Simulation in Developing Student Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Juliana de Lima Lopes, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 43095115.9.0000.5505
Record Dates: First submitted 2017-10-02; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Students
Keywords: students, nursing; simulation training; Instructional Films and Videos; Aptitude

STUDY DESIGN:
Intervention Model Description: The students were randomized to one of two groups (control or intervention), according to the sequence determined by the Random System
Who Masked: Investigator, Outcomes Assessor
Masking Description: The teacher that evaluated the students, was not informed if the student was of the control or intervention group. The outcomes assessor was not informed if the group 1 and 2 was control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video during simulation (Experimental): The intervention group simulated the bed bath while watching the video, under the supervision of the tutor
  Interventions: Other: Video during simulation
- Simulation without video (No Intervention): The students of the control group performed the simulation of the bed bath procedure, with the aid of a tutor.

INTERVENTIONS:
Other: Video during simulation — The intervention group simulated the bed bath while watching the video, under the supervision of the tutor
  Other Names: Educational
  Arms: Video during simulation

SUMMARY:
This study´s objective was to identify the effectiveness of bed bath video during simulation in the performance of undergraduate student skills. Method. This is a randomized, blinded clinical trial. The sample consisted of students of the second year of nursing graduation who were divided into two groups: intervention group (students who simulated bed bath using the video) and control group (students who simulated bed bath without the video). The primary end point was the performance of the students' abilities about bed bath procedure, which was evaluated in two moments (before and after the simulation) and we used a previously elaborated and validated checklist. Prior to the collection, the research project was submitted to the Research Ethics Committee and the data was collected after its approval.

DETAILED DESCRIPTION:
This study´s objective was to identify the effectiveness of bed bath video during simulation in the performance of undergraduate student skills. Method. This is a randomized, blinded clinical trial. The sample consisted of students of the second year of nursing graduation who were divided into two groups: intervention group (students who simulated bed bath using the video) and control group (students who simulated bed bath without the video). The students attended an expository dialog class about bed bath, structured on the basis of literature and that subsidized the elaboration of the video and the instrument to evaluate of the performance of the abilities. After the class, the subjects were consulted about the desire to participate, and those who agreed, signed the consent form. After the theoretical class, students were invited to attend the UNIFESP Skills and Simulation Teaching Center and were randomized to one of two groups (control or intervention), according to the sequence determined by the Random System. Randomization was carried out by a teacher who did not participate of any phase of this study, with masking of this phase. After randomization, the student was instructed to perform the bed bathing procedure on the low fidelity manikin, based on the knowledge obtained in the theoretical class, and no guidance was given at this time. At this stage, the teacher evaluated the student's skills through the checklist. It is emphasized that this teacher was not informed if the student evaluated was of the control group or intervention, and there is masking of this phase. The instrument for evaluating the performance of bed bath skills was the previously prepared and validated checklist called "Instrument for bathing in the bed - IABL", which presented good internal consistency in the validation study (Cronbach's alpha = 0.896) . This instrument is composed of three topics (nursing orientation, material preparation and procedure) and 56 items, whose scores vary from 0 to 56 points, in which the higher the score the better the students' abilities performance. Each item of this instrument was observed during the execution of the procedure before and after the simulation and was considered as executed properly (1 point), inadequate (0 point) or not performed (0 point). The performance of each student was analyzed by adding the scores of the items of the instrument. Subsequent to this first evaluation, the students, both in the control group and in the intervention group, received the intervention by another teacher. The students of the control group performed the simulation of the bed bath procedure, with the aid of a tutor and the intervention group simulated the bed bath while watching the video, under the supervision of the tutor. The tutor, from both groups, acted as facilitator of the teaching-learning process, according to the needs presented during the simulation period. At the end of the simulation, the student of both groups was instructed to perform the bed bath procedure once again, and no guidance was given at this time. The performance of the student's abilities was evaluated by the same instrument and by the same teacher of the first evaluation. Prior to the collection, the research project was submitted to the Research Ethics Committee and the data was collected after its approval.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years

Exclusion Criteria:

* Students who have ever performed the bed bath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2016-03-08 (Actual)

PRIMARY OUTCOMES:
Change from score of student's skills about bed bath | The students were followed for two days
  The student's skills was evaluated using the checklist previously elaborated and validated, immediately before and after interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana de Lima Lopes, PhD, Principal Investigator — Federal University of São Paulo; Alba LB Barros, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We not plan to make individual participant data avaiable to other researchers.

REFERENCES:
- [Background] Baxter P, Akhtar-Danesh N, Valaitis R, Stanyon W, Sproul S. Simulated experiences: nursing students share their perspectives. Nurse Educ Today. 2009 Nov;29(8):859-66. doi: 10.1016/j.nedt.2009.05.003. Epub 2009 Jun 4. PMID 19500886
- [Background] Fleming SE, Reynolds J, Wallace B. Lights... camera... action! a guide for creating a DVD/video. Nurse Educ. 2009 May-Jun;34(3):118-21. doi: 10.1097/NNE.0b013e3181a0270e. PMID 19412052